CLINICAL TRIAL: NCT05371431
Title: The Effect of Individualized Blood Flow Restriction Training on the Patients Following the Conservative Treatment of Distal Radius Fracture
Brief Title: The Effect of Blood Flow Restriction Training on the Patients of Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY20200820-01
Record Dates: First submitted 2022-04-06; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-BFR groups (Experimental): Traditional rehabilitation training is designed according to postoperative orthopaedic rehabilitation guidelines. Traditional rehabilitation trainings include grip and pinch, wrist flexion with forearm pronated, wrist extension with forearm pronated, wrist flexion with forearm supinated, wrist extension with forearm supinated, prayer sign (wrist flexion), prayer sign (wrist extension), forearm pronation, forearm supination. Patients participated in 2 training sessions per week with at least 48 hours rest in between for continuous 6 weeks.
  Interventions: Other: Traditional rehabilitation training
- BFR groups (Experimental): Patients in the BFR group underwent the same traditional rehabilitation training protocol with non-BFR utilizing a medical grade tourniquet system (ATS 4000 TS，Zimmer Surgical, Inc. Dover). The ATS 4000 tourniquet system tailors the individualized tourniquet pressure to each patient following determination of the limb occlusion pressure (LOP), and studies have shown that 50% LOP is safe and effective in the rehabilitation of DRF. When the tourniquet system was used, LOPs were reassessed for every session before training, and pressures were continually monitored. Participants were to perform the entirety of each training (including intra-set rest periods) under 50% LOP with the tourniquets released during the 2-minute rest periods between sets. Patients participated in 2 training sessions per week with at least 48 hours rest in between for continuous 6 weeks.
  Interventions: Other: Blood flow restriction combined with traditional rehabilitation training

INTERVENTIONS:
Other: Traditional rehabilitation training — The non-BFR group undertook traditional rehabilitation training only. Patients participated in 2 training sessions per week with at least 48 hours rest in between for continuous 6 weeks. Clinical assessment of grip strength, pinch strength (tip pinch strength, key pinch strength and tripod pinch strength), ROM of wrist, PRWE score, muscle stiffness and radiographic outcomes, was conducted at the 6th and 12th week from the date of initial DRF.
  Arms: non-BFR groups
Other: Blood flow restriction combined with traditional rehabilitation training — BFR group completed the traditional rehabilitation training with a medical grade tourniquet applied on the upper arm. Patients participated in 2 training sessions per week with at least 48 hours rest in between for continuous 6 weeks. Clinical assessment of grip strength, pinch strength (tip pinch strength, key pinch strength and tripod pinch strength), ROM of wrist, PRWE score, muscle stiffness and radiographic outcomes, was conducted at the 6th and 12th week from the date of initial DRF.
  Arms: BFR groups

SUMMARY:
The aim of this study was to compare the effect of blood flow restriction (BFR) training and traditional rehabilitation training on grip strength, pinch strength (tip pinch strength, key pinch strength and tripod pinch strength), range of motion (ROM) of wrist, patient-rated wrist evaluation (PRWE) score, muscle stiffness and radiographic outcomes in distal radius fracture (DRF) patients during a post-treatment rehabilitation program.

DETAILED DESCRIPTION:
This study is a randomized controlled study. Patients in the non-BFR group underwent a traditional rehabilitation training. Traditional rehabilitation training is designed based on post injury rehabilitation guidelines. This guideline recommends that the early rehabilitation of DRF should be progressive, with training loads ranging from self-weight to full weight bearing depending on the patient's individual situation. During the six weeks, a progressive training load has been applied to the patients. First week: no weight bearing. Second to sixth week: resistance was increased by 1LB (~0.45 kg) for individual training only if a participant could consecutively achieve at least 30/15/15/15 (75 total) repetitions for both training sessions within a given training week. The exercises include grip and pinch, wrist flexion with forearm pronated, wrist extension with forearm pronated, wrist flexion with forearm supinated, wrist extension with forearm supinated, prayer sign (wrist flexion), prayer sign (wrist extension), forearm pronation, and forearm supination. Patients participated in 2 training sessions per week with at least 48 hours rest in between for continuous 6 weeks. BFR training twice a week for at least 6 weeks has been reported to increase muscle hypertrophy and strength. The BFR group underwent the same traditional rehabilitation training program but combined with BFR implemented by a medical grade tourniquet system (ATS 4000 TS，Zimmer Surgical, Inc. Dover). The tourniquet system consists of a ATS 4000 tourniquet system, and a tourniquet cuff (10 cm × 46 cm). The ATS 4000 tourniquet system tailors the individualized tourniquet pressure to each patient following determination of the limb occlusion pressure (LOP), and studies have shown that 50% LOP is safe and effective in the rehabilitation of DRF. When the tourniquet system was used, LOPs were reassessed for every session before training, and pressures were continually monitored. Participants were to perform the entirety of each training (including intra-set rest periods) under 50% LOP with the tourniquets released during the 2-minute rest periods between sets.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 75 years
* Colles' fracture
* No history of wrist injury or joint deformity
* No other types of upper limb injuries occurred in the last 3 months
* No cardiovascular diseases

Exclusion Criteria:

* Concurrent ipsilateral upper limb fracture
* Concurrent bilateral upper limb fractures
* History of surgery or any invasive procedure on the upper limb
* History of peripheral arterial disease or deep vein thrombosis
* History of cancer that has generated limitations or restrictions to physical exercise

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
grip strength | Conducted at the 6th week from the date of initial gypsum immobilization.
  Grip strength (JA Preston, Corporation Jackson, MI, USA) was measured in method recommended by the American Society of Hand Therapists. The scale of the dynamometer indicated handgrip strength in kilograms (kg). The testing protocol consisted of three maximal voluntary isometric contractions maintained for 5 s, with rest period of at least 60 s; the highest value was used for the determination of the maximal grip strength. Participants standing, shoulder in a neutral position, arm by side, elbow fully extended. Specific verbal instructions were given to subjects before the evaluations and the experiments were performed with verbal encouragement.
grip strength | Conducted at the 12th week from the date of initial gypsum immobilization.
  Grip strength (JA Preston, Corporation Jackson, MI, USA) was measured in method recommended by the American Society of Hand Therapists. The scale of the dynamometer indicated handgrip strength in kilograms (kg). The testing protocol consisted of three maximal voluntary isometric contractions maintained for 5 s, with rest period of at least 60 s; the highest value was used for the determination of the maximal grip strength. Participants standing, shoulder in a neutral position, arm by side, elbow fully extended. Specific verbal instructions were given to subjects before the evaluations and the experiments were performed with verbal encouragement.
Pinch Strength | Conducted at the 6th week from the date of initial gypsum immobilization.
  Pinch strength (B&L Engineering, Sana Ana, CA) were measured in method recommended by the American Society of Hand Therapists. Participants were seated with their shoulder adducted and neutrally rotated, elbow flexed to 90°, forearm in neutral position. Three measurements were made and the average value was used.
Pinch Strength | Conducted at the 12th week from the date of initial gypsum immobilization.
  Pinch strength (B&L Engineering, Sana Ana, CA) were measured in method recommended by the American Society of Hand Therapists. Participants were seated with their shoulder adducted and neutrally rotated, elbow flexed to 90°, forearm in neutral position. Three measurements were made and the average value was used.
ROM of the wrist | Conducted at the 6th week from the date of initial gypsum immobilization.
  ROM of the wrist (wrist flexion, extension, radial deviation, ulnar deviation; forearm supination and pronation) was measured by a goniometer in positions recommended by the American Society of Hand Therapists. Three measurements were made and the average value was used.
ROM of the wrist | Conducted at the 12th week from the date of initial gypsum immobilization.
  ROM of the wrist (wrist flexion, extension, radial deviation, ulnar deviation; forearm supination and pronation) was measured by a goniometer in positions recommended by the American Society of Hand Therapists. Three measurements were made and the average value was used.
PRWE Score | Conducted at the 6th week from the date of initial gypsum immobilization.
  The PRWE is a region specific outcome measure that evaluates wrist-related disability. It contains 15 items: five of which evaluate pain (intensity and frequency) and 10 evaluate function (specific activities and usual activities). Participants are instructed to answer all questions by rating their average pain and level of function over the past week. To produce the function subscale score, the responses to the 10 functional items are tallied and divided by two. Adding the pain and function subscale scores produces the total PRWE score, where 0 is the best score (no pain or difficulty performing activities) and 100 is the worse score (severe continuous pain and unable to perform activities).
PRWE Score | Conducted at the 12th week from the date of initial gypsum immobilization.
  The PRWE is a region specific outcome measure that evaluates wrist-related disability. It contains 15 items: five of which evaluate pain (intensity and frequency) and 10 evaluate function (specific activities and usual activities). Participants are instructed to answer all questions by rating their average pain and level of function over the past week. To produce the function subscale score, the responses to the 10 functional items are tallied and divided by two. Adding the pain and function subscale scores produces the total PRWE score, where 0 is the best score (no pain or difficulty performing activities) and 100 is the worse score (severe continuous pain and unable to perform activities).
Muscle Stiffness | Conducted at the 6th week from the date of initial gypsum immobilization.
  Muscle stiffness (MyotonPRO, Myoton Ltd, Estonia) was measured in method recommended by the Ditroilo et al. Participants were required to expose their arms in the relaxed position. To maintain consistency of measurements among participants, marks were drawn on the skin in the following site on arm. Five consecutive measurements were taken. The average of the five measurements was used for later analysis.
Muscle Stiffness | Conducted at the 12th week from the date of initial gypsum immobilization.
  Muscle stiffness (MyotonPRO, Myoton Ltd, Estonia) was measured in method recommended by the Ditroilo et al. Participants were required to expose their arms in the relaxed position. To maintain consistency of measurements among participants, marks were drawn on the skin in the following site on arm. Five consecutive measurements were taken. The average of the five measurements was used for later analysis.

SECONDARY OUTCOMES:
Radiographic outcomes | Conducted at 1th week(post injury).
  Anteroposterior and lateral radiographs (Kodak DR, DR Evolution, Eastman Kodak) were acquired at pre and post training as safety indicators. Radiographic outcomes were measured by doctors of the same profession.
Radiographic outcomes | Conducted at 1th week(post reduction).
  Anteroposterior and lateral radiographs (Kodak DR, DR Evolution, Eastman Kodak) were acquired at pre and post training as safety indicators. Radiographic outcomes were measured by doctors of the same profession.
Radiographic outcomes | Conducted at 6th week.
  Anteroposterior and lateral radiographs (Kodak DR, DR Evolution, Eastman Kodak) were acquired at pre and post training as safety indicators. Radiographic outcomes were measured by doctors of the same profession.
Radiographic outcomes | Conducted at 12th week.
  Anteroposterior and lateral radiographs (Kodak DR, DR Evolution, Eastman Kodak) were acquired at pre and post training as safety indicators. Radiographic outcomes were measured by doctors of the same profession.

CONTACTS AND LOCATIONS:
Overall Officials: bin Liang, Prof, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Yang M, Liang B, Zhao X, Wang Y, Xue M, Song Q, Wang D. The effectiveness of individualized blood flow restriction training following patellar fracture surgery: a case series. BMC Musculoskelet Disord. 2025 Mar 12;26(1):247. doi: 10.1186/s12891-025-08424-2. PMID 40075367
- [Derived] Yang M, Liang B, Zhao X, Wang Y, Xue M, Wang D. BFR Training Improves Patients' Reported Outcomes, Strength, and Range of Motion After Casting for Colles' Fracture. Med Sci Sports Exerc. 2023 Nov 1;55(11):1985-1994. doi: 10.1249/MSS.0000000000003228. Epub 2023 Jun 1. PMID 37259253